CLINICAL TRIAL: NCT00042081
Title: A Phase III, Multi-Center Randomized, Double-Blind, Placebo-Controlled Trial of the Ex Vivo Treatment With CGT003 of Coronary Vein Grafts in Patients Undergoing Coronary Artery Bypass Graft Procedures
Brief Title: Prevention of Autogenous Vein Graft Failure in Coronary Artery Bypass Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anesiva, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CGT003-04
Record Dates: First submitted 2002-07-22; First posted 2002-07-24 (Estimated); Last update posted 2006-05-05 (Estimated); Status verified 2005-07

CONDITIONS: Coronary Artery Disease
Keywords: CABG; coronary artery bypass surgery; coronary artery disease; coronary arteriosclerosis; coronary stenosis; coronary occlusion
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Coronary Occlusion

INTERVENTIONS:
Drug: CGT003 (E2F Duplex Decoy)

SUMMARY:
The purpose of this study is to determine the efficacy of graft pretreatment with CGT003 (E2F Duplex Decoy), as compared to placebo, on the incidence of patients experiencing vein graft failure after coronary artery bypass surgery.

DETAILED DESCRIPTION:
Coronary vascular disease manifested by narrowing of the coronary arteries is one of the more common manifestations of atherosclerotic vascular disease. The clinical manifestations of coronary artery disease include death, angina pectoris, myocardial infarction, congestive heart failure and arrhythmia. Restoration of circulation to the heart may be undertaken using a variety of techniques including angioplasty, stenting, and bypass grafting.

Approximately 359,000 patients underwent coronary bypass procedures in the U.S. in 1999. Long term studies have observed an incidence of vein graft occlusion at 19% at 1 year, 25% at 5 years and 50% by 15 years after operation for an overall rate of 2.5% per year after the first year of observation. The consequences of graft failure are as significant as those of primary atherosclerotic disease and include ischemia, myocardial infarction and death.

CGT003 is a novel therapeutic that is under investigation as a treatment to prevent vein graft failure. It acts by inhibiting the transcription factor, E2F, which is activated in response to injury such as that which occurs when thin-walled vein grafts are exposed to the pressures of the arterial circulation. Blockade of E2F inhibits smooth muscle cell proliferation and redirects the vein graft remodeling that occurs within the first several days after implantation towards medial hypertrophy and strengthening of the medial layer and blunts formation of neointima. Inhibition of neotinimal formation coupled with expansion of the media should result in a decreased risk of the accelerated atherosclerosis and consequent vein graft failure over several years.

ELIGIBILITY:
PATIENTS MUST:

* Have coronary artery disease and be scheduled to undergo a coronary artery bypass (CABG) procedure that is to include at least two segments of autogenous vein (sequential grafts do not count as two separate grafts).
* Be between 18 and 80 years old.
* Have a documented negative serum pregnancy test for all women of childbearing potential.
* Be using an acceptable method of birth control if of reproductive potential.
* Have agreed to participate voluntarily and signed and dated an IRB-approved, Patient Informed Consent form.
* (If one of the first 2400 patients enrolled) have agreed to participate voluntarily and signed and dated an IRB-approved, Patient Informed Consent form for the Angiography population.
* Note: Patients who are to receive an arterial bypass to the left anterior descending artery in addition to the two vein grafts required by the protocol ARE eligible for this study.
* Note: Patients ARE eligible for enrollment regardless of whether the planned procedure is to be on or off cardiopulmonary bypass pump.
* Note: Patients who do not wish to undergo elective Angiography at one year SHOULD NOT be enrolled in the first 2400 patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000
Dates: Start 2002-07; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: Todd Lorenz, M.D., Study Director — Anesiva, Inc.
Locations (152):
- United States (152):
  - Brookwood Medical Center, Birmingham, Alabama
  - Cardio-Thoracic Surgeons, P.C., Birmingham, Alabama
  - Baptist Medical Center - Montclair, Birmingham, Alabama
  - Medical Center East, Birmingham, Alabama
  - Seton Medical Center, Daly City, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Desert Regional Medical Center, Palm Springs, California
  - St. Joseph's Medical Center, Stockton, California
  - St. Vincent's Medical Center, Bridgeport, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Cardiovascular Research, Atlantis, Florida
  - JFK Medical Center, Atlantis, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - Cardiovascular Surgeons, P.A., Orlando, Florida
  - Florida Hospital, Orlando, Florida
  - Orlando Cardiovascular Center, LLLP, Orlando, Florida
  - Orlando Heart Center, Orlando, Florida
  - Orlando Regional Med Center, Orlando, Florida
  - Orlando Heart Center/Sand Lake, Orlando, Florida
  - Clinical Research Center, Sarasota, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Crawford Long Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - St. Elizabeth's Hospital, Belleville, Illinois
  - Memorial Hospital, Belleville, Illinois
  - Northwestern Medical Facility Foundation, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Rush Professional Building, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Evanston Northwestern Healthcare, Highland Park Hospital, Evanston, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - St. Francis Hospital of Evanston, Evanston, Illinois
  - Loyola University Chicago Medical Center, Maywood, Illinois
  - Edward Hospital & Health Services, Naperville, Illinois
  - Advocate Christ Hospital and Medical Center, Oak Lawn, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Dep. of Surgery, Div. of Cardiothoracic Surgery, Springfield, Illinois
  - Southern Illinois University School of Medicine, Department of Surgery, Division of Cardiothoracic Surgery, Springfield, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - St. Vincent Hospital and Health Care Service, Indianapolis, Indiana
  - The Heart Center of Indiana, Indianapolis, Indiana
  - Genesis Heart Institute, Davenport, Iowa
  - Genesis Medical Center, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Georgetown Professional Plaza, Overland Park, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Jewish Hospital Health Care Services, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Cardiac Surgery Associates, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Cardiac Surgery Associates, Towson, Maryland
  - Midatlantic Cardiovascular Associates, P.A., Towson, Maryland
  - St. Joseph Medical Center, Towson, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - McLaren Regional Medical Center, Flint, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Ingham Regional Medical Center, Lansing, Michigan
  - Thoracic & Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Thoracic & Cardiovascular Institute, Lansing, Michigan
  - Cardiology Consultants, PC, Petoskey, Michigan
  - Great Lakes Cardiothoracic and Vascular Surgery, Petoskey, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Petoskey Cardiology, Petoskey, Michigan
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - Convenant Medical Center, Saginaw, Michigan
  - St. Mary's/Duluth Clinic Health System, Duluth, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Institute, Minneapolis, Minnesota
  - Methodist Hospital, Saint Louis Park, Minnesota
  - Park Nicollet Heart Center, Saint Louis Park, Minnesota
  - Forrest General Hospital, Hattiesburg, Mississippi
  - St. John's Regional Medical Center, Joplin, Missouri
  - 930 Carondelet Drive, Kansas City, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nebraska Heart Institute, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nebraska Heart Institute, Papillion, Nebraska
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Umdnj-Rwjms, New Brunswick, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Lenox Hill Hospital, New York, New York
  - New York Presbyterian Medical Center, Milstein Hospital Building, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Ambulatory Care Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - Brody School of Medicine, East Carolina University, Greenville, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Forysyth Medical Center, Winston-Salem, North Carolina
  - Walley, Morgan & Duncan, M.D., P.A., Winston-Salem, North Carolina
  - MeritCare Clinic at MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Cardiovascular & Thoracic Surgeons, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Cardiovascular & Thoracic Surgeons, Inc., Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Kettering Medical Center Network, Kettering Hospital, Kettering, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Presbyterian Hospital, University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Guthrie Clinic, Sayre, Pennsylvania
  - Robert Packer Hospital, Sayre, Pennsylvania
  - The Chester County Hospital, West Chester, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Upstate Cardiothoracic Surgery, Greenville Hospital System, Greenville, South Carolina
  - Saint Francis Hospital, Memphis, Tennessee
  - Heart Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - St. Paul University Hospital, Dallas, Texas
  - Denton Regional Medical Center, Denton, Texas
  - Medical Center Plano, Plano, Texas
  - Southwest Texas Methodist Hospital, San Antonio, Texas
  - Northeast Methodist Hospital, San Antonio, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Lynchburg General Hospital, Lynchburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Mid-Atlantic Cardiothoracic Surgeons, Ltd., Norfolk, Virginia
  - St. Joseph Hospital, Bellingham, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Northwest Heart and Lung Surgical Associates, Spokane, Washington
  - CAMC Health Education and Research Institute, Clinical Trials Center, Charleston, West Virginia
  - Charleston Area Medical Center, Charleston, West Virginia
  - Appleton Heart Institute at Appleton Medical Center, Appleton, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Community Health Care/Wausau Hospital, Wausau, Wisconsin
  - Wausau Heart and Lung Surgeons, Wausau, Wisconsin

REFERENCES:
- [Result] Alexander JH, Hafley G, Harrington RA, Peterson ED, Ferguson TB Jr, Lorenz TJ, Goyal A, Gibson M, Mack MJ, Gennevois D, Califf RM, Kouchoukos NT; PREVENT IV Investigators. Efficacy and safety of edifoligide, an E2F transcription factor decoy, for prevention of vein graft failure following coronary artery bypass graft surgery: PREVENT IV: a randomized controlled trial. JAMA. 2005 Nov 16;294(19):2446-54. doi: 10.1001/jama.294.19.2446. PMID 16287955
- [Derived] Harskamp RE, Alexander JH, Ferguson TB Jr, Hager R, Mack MJ, Englum B, Wojdyla D, Schulte PJ, Kouchoukos NT, de Winter RJ, Gibson CM, Peterson ED, Harrington RA, Smith PK, Lopes RD. Frequency and Predictors of Internal Mammary Artery Graft Failure and Subsequent Clinical Outcomes: Insights From the Project of Ex-vivo Vein Graft Engineering via Transfection (PREVENT) IV Trial. Circulation. 2016 Jan 12;133(2):131-8. doi: 10.1161/CIRCULATIONAHA.115.015549. Epub 2015 Dec 8. PMID 26647082
- [Derived] Hess CN, Lopes RD, Gibson CM, Hager R, Wojdyla DM, Englum BR, Mack MJ, Califf RM, Kouchoukos NT, Peterson ED, Alexander JH. Saphenous vein graft failure after coronary artery bypass surgery: insights from PREVENT IV. Circulation. 2014 Oct 21;130(17):1445-51. doi: 10.1161/CIRCULATIONAHA.113.008193. Epub 2014 Sep 26. PMID 25261549
- [Derived] Harskamp RE, Alexander JH, Schulte PJ, Brophy CM, Mack MJ, Peterson ED, Williams JB, Gibson CM, Califf RM, Kouchoukos NT, Harrington RA, Ferguson TB Jr, Lopes RD. Vein graft preservation solutions, patency, and outcomes after coronary artery bypass graft surgery: follow-up from the PREVENT IV randomized clinical trial. JAMA Surg. 2014 Aug;149(8):798-805. doi: 10.1001/jamasurg.2014.87. PMID 25073921
- [Derived] Lopes RD, Williams JB, Mehta RH, Reyes EM, Hafley GE, Allen KB, Mack MJ, Peterson ED, Harrington RA, Gibson CM, Califf RM, Kouchoukos NT, Ferguson TB, Lorenz TJ, Alexander JH. Edifoligide and long-term outcomes after coronary artery bypass grafting: PRoject of Ex-vivo Vein graft ENgineering via Transfection IV (PREVENT IV) 5-year results. Am Heart J. 2012 Sep;164(3):379-386.e1. doi: 10.1016/j.ahj.2012.05.019. PMID 22980305